CLINICAL TRIAL: NCT06218524
Title: Clinical Study for Evaluating the Effectiveness of Haloperidol and Temozolomide Synergism on Adult Recurrence Glioblastoma
Brief Title: The Effectiveness of HP and TMZ Synergism on Adult Recurrence GBM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Yuntao Lu, Professor, Neurosurgeon, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEC-DRD2
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Chemoresistance; Autophagy; Ferropotosis; DRD2; Haloperidol
MeSH Terms: conditions — Glioblastoma | interventions — Haloperidol; Temozolomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMZ single (Placebo Comparator): Single oral Temozolomide
  Interventions: Drug: Temozolomide
- TMZ and Haloperidol (Experimental): Oral Temozolomide and Haloperidol
  Interventions: Drug: Haloperidol Tablets; Drug: Temozolomide

INTERVENTIONS:
Drug: Haloperidol Tablets — Haloperidol tablet 6mg, Oral, Triple/Day
  Arms: TMZ and Haloperidol
Drug: Temozolomide — Temozolomide, 150mg/kg, Oral, Once/Day, 5/28 days

SUMMARY:
The study of investigators indicated that TMZ can up-regulate dopamine D2 receptor (DRD2) expression, and mediates Ferroptosis inhibition and chemoresistance of GBM. The clinical data also proved that the DRD2 expression in recurrent GBM is significantly higher than that in primary GBM. Moreover, the DRD2 antagonist haloperidol can attenuate the above function of DRD2, and increase the sensitivity of GBM to the TMZ by inducing fatal autophagy and ferroptosis. In xenograft mice, the combined usage of haloperidol and Temozolomide (TMZ) can significantly inhibit tumor growth and increase overall survival. The investigators' findings have been published in Clinical cancer research. Haloperidol known as a butylbenzene antipsychotic drug, has been widely used in several kinds of mental illnesses, such as depression, schizophrenia, and Bipolar disorder. And the safe dosage of the haloperidol is clear so far. So in this study, the investigators will recruit the patients who suffered from recurrent GBM, and evaluate the effectiveness of single TMZ chemotherapy or combined with haloperidol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Primary GBM underwent surgery and TMZ chemoradiotherapy, and MRI confirmed the tumor recurrence
* Without severe cardiac diseases

Exclusion Criteria:

* Child patients (<18 years)
* Recurrence tumors grow fast, which needs surgery removal
* H3K27M midline glioblastoma
* Suffered with severe cardiac diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of partial relief and complete relief | 3 months
  Detected the percentage of partial relief and complete relief according to RANO criteria.

SECONDARY OUTCOMES:
Overall survival | One year
  Overall survival was evaluated during follow-up period.
DRD2 expression | One year
  If the recurrent GBM underwent surgery resection, the DRD2 expression was detected.

OTHER OUTCOMES:
Adverse drug reaction of haloperidol | One year
  Detection the adverse drug reaction of haloperidol

CONTACTS AND LOCATIONS:
Overall Officials: Yuntao Lu, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Result] Shi L, Chen H, Chen K, Zhong C, Song C, Huang Y, Wang T, Chen L, Li C, Huang A, Qi S, Li H, Lu Y. The DRD2 Antagonist Haloperidol Mediates Autophagy-Induced Ferroptosis to Increase Temozolomide Sensitivity by Promoting Endoplasmic Reticulum Stress in Glioblastoma. Clin Cancer Res. 2023 Aug 15;29(16):3172-3188. doi: 10.1158/1078-0432.CCR-22-3971. PMID 37249604
- See also: Our study about the anti-tumor function of Haloperidol, which was published in Clinical Cancer research. — https://pubmed.ncbi.nlm.nih.gov/37249604/